CLINICAL TRIAL: NCT05864651
Title: Tele-Exercise Programs Improves Physical Performance for Male Elite Fencers
Brief Title: Tele-Exercise for Male Elite Fencers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Sungbae Jo, Physical Therapist, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SYU 2022-10-015-001
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Sports Physical Therapy; Athletic Performance
Keywords: Sports Physical Therapy; Athletic Performance; Fencing; Tele-exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-exercise program group (Experimental): Provide the following programs:
  1. tele-exercise program: 5 times per week, 30 minute/session
  2. conventional fencing exercise: 5 times per week, 30 minute/session
  Interventions: Other: Tele-exercise program; Other: Conventional Fencing Exercise
- Control group (Active Comparator): Provide the following programs:
  1) conventional fencing exercise: 5 times per week, 30 minute/session
  Interventions: Other: Conventional Fencing Exercise

INTERVENTIONS:
Other: Tele-exercise program — The tele-exercise program focused on lunge movement with additional strengthening abdominal and lumbopelvic muscle training while maintaining neuromuscular control. The difficulty of training was adjusted every week according to the five-step mastery program
  Arms: Tele-exercise program group
Other: Conventional Fencing Exercise — The conventional exercise was based on 'displacement', a basic footwork training in fencing. The Displacement is also basic footwork to approach the opponent. The Displacement consisted of seven movements including 'Marche', 'Retraite & Rompre', 'Passe avant', 'Passe arrière', 'Bond en avant', 'Bond en arrière', and 'Balestra'.

SUMMARY:
Tele-exercise has been used to enhance athletic performance among athletes. Physical performance indicators such as lunge distance, speed, reaction time, coordination, and balance control during stationary jumps can be used to measure the effectiveness of tele-exercise programs for fencing athletes.

The objective of this study was to examine the effectiveness of tele-exercise programs on lunge distance, speed, reaction time, coordination, and balance control during stationary jumps among male elite fencers.

ELIGIBILITY:
Inclusion Criteria:

* who are registered to Elite Fencer to both Korean Sports & Olympic Committee and Korean Fencing Federation;
* who does not have a history of musculoskeletal or neurological injuries in the past six months;
* who have no physical limitations.

Exclusion Criteria:

* Those who have the experience of participating in experiments in the past year
* who refuses to participate or provide written consent.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Lunge speed | changes from baseline after intervention at 4 weeks
  Speed to perform a single lunge is one of the essential physical ability for fencing athletes.
Lunge distance | changes from baseline after intervention at 4 weeks
  Distance travelled to perform a single lunge is one of the essential physical ability for fencing athletes.
Reaction time | changes from baseline after intervention at 4 weeks
  Reaction time is one of the essential physical ability for fencing athletes that can be measured by the time required to move when subject hear a signal

SECONDARY OUTCOMES:
Accurate repeatability of stationary hops | changes from baseline after intervention at 4 weeks
  The distances between repeated hops can evaluate coordination and balance control

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physicla Therapy, Sahmyook University, Seoul, South Korea